CLINICAL TRIAL: NCT05455151
Title: Hysteroscopic Injections of Autologous Endometrial Cells and Platelet-rich Plasma in Patients With Thin Endometrium - a Pilot Study
Brief Title: Hysteroscopic Injections of Autologous Endometrial Cells and Platelet-rich Plasma in Patients With Thin Endometrium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Collaborators: Sechenov University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: №10-18/11.2018
Record Dates: First submitted 2022-06-28; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Thin Endometrium
Keywords: platelet-rich plasma; infertility; endometrial cells
MeSH Terms: conditions — Infertility | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: The patients were divided into 4 groups depending on the substances introduced into the basal layer of the endometrium. Group 1 underwent conservative therapy. Group 2 received intraendometrial injections of autologous PRP instead of the conservative therapy. Group 3 received identical injections after conservative therapy. Group 4 received injections of the minimally manipulated autologous endometrial cells suspended in autologous PRP.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conservative therapy (Active Comparator): This is Group 1, whose patients received electrical impulse therapy using a BTL-4000 Premium G device (BTL Medical Technologies, Czech Republic) starting from day 5-7 of menstrual cycle for 10-12 days daily.
  Interventions: Procedure: Conservative therapy
- PRP injection (Experimental): This is Group 2, whose patients received single intraendometrial injections of autologous PRP during proliferative phase (day 6-9) of menstrual cycle.
  Interventions: Biological: PRP injection
- Injection of PRP after conservative therapy (Experimental): This is Group 3, whose patients received electrical impulse therapy identically with Group 1 during the first menstrual cycle. In the second cycle, the patients received autologous PRP injections identically with Group 2.
  Interventions: Biological: Injection of PRP after conservative therapy
- Injection of PRP with endometrial cells (Experimental): This is Group 4, whose patients received single intraendometrial injections of the minimally manipulated autologous endometrial cells suspended in autologous PRP during proliferative phase (day 6-9) of menstrual cycle.
  Interventions: Biological: Injection of PRP with endometrial cells

INTERVENTIONS:
Procedure: Conservative therapy — Conservative therapy to which the patients were subjected was the effect of an electrical impulse
  Arms: Conservative therapy
Biological: PRP injection — This intervention consisted of injecting platelet-rich plasma (PRP) into the endometrium
  Arms: PRP injection
Biological: Injection of PRP after conservative therapy — This intervention consisted of conducting conservative therapy with an electrical impulse and then injecting PRP inside the endometrium
  Arms: Injection of PRP after conservative therapy
Biological: Injection of PRP with endometrial cells — This intervention consisted of injecting endometrial cells suspended in prp
  Arms: Injection of PRP with endometrial cells

SUMMARY:
The investigation is devoted to the study of the effect of the introduction of autologous platelet-rich plasma (PRP) on the thickness of the endometrium. It was found that the injection of PRP and endometrial cells resuspended in PRP into the endometrium of patients with thin endometrium leads to an increase in the proliferation of endometrial cells, and as a result, to an increase in its thickness.

DETAILED DESCRIPTION:
The study enrolled 115 patients with thin endometrium (<7 mm at implantation window) and infertility. The cohort was divided into groups based on the treatment regimen.

Group 1 (the control, n=30) underwent conservative therapy. Group 2 (n=42) received intraendometrial injections of autologous PRP instead of the conservative therapy. Group 3 (n=38) received identical injections after conservative therapy. Group 4 (n=5) received injections of the minimally manipulated autologous endometrial cells suspended in autologous PRP.

Injections of PRP and endometrial cells suspended in autologous PRP into basal layer of endometrium facilitate the reconstitution by enhancing cell proliferation and angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Normal karyotype
* Normal karyotype of the partner
* Regular ovulatory and menstrual cycle
* Endometrium <7 mm thick as measured at implantation window
* Availability of ≥2 vitrified blastocysts of good quality
* History of implantation failure and/or embryo transfer (ET) cancellation due to insufficient endometrial thickness

Exclusion Criteria:

* Pathospermia in partner
* Use of donor gametes
* Premature ovarian failure
* Internal genital anomalies
* Systemic blood diseases and coagulopathy
* Hemoglobin <100 g/L
* Platelets <100×109/L
* Antiplatelet/anticoagulant therapy recipient status

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 115 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in endometrial thickness after treatment compared with control. | Baseline and 2 month
  Ultrasonography measurements of endometrial thickness before and after the therapy and compare the thickness. Endometrial thickness measured in mm.
The Doppler-assisted detection of the uterine spiral arteries | 1 month
  The number of identified vessels is counted and the percentage of detection frequency is calculated accordingly, adjusted for the McNemar's binomial test. Compare the rates of visualization of the uterine spiral arteries after therapy in all groups of patients.
Study of the effect of therapy on the onset of pregnancy | 9 months
  Investigation of the rates of clinical pregnancies and live births in all groups. After therapy, the number of clinical pregnancy and the number of live births were calculated.
The content of growth factor in autologous PRP | 3 month
  Investigation of the content of platelet-derived growth factor-BB (PDGF-BB) and vascular endothelial growth factor (VEGF) in autologous PRP. Relative levels of PDGF-BB and VEGF are normalized to the total protein content.
Phenotyping of cells isolated from endometrial biopsies | 3 month
  Investigation of cellular composition in endometrial biopsy. The percentage of cells positive for markers of mesenzymal stromal cells, epithelial and endothelial cells, lymphocytes is calculated and the determination of the phenotype of cells in endometrial biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Inna Apolikhina, MD, Study Director — FSBI "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov" Ministry of Healthcare of the Russian Federation; Zulfiia Efendieva, PhD, Principal Investigator — FSBI "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov" Ministry of Healthcare of the Russian Federation
Locations (1):
- Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow, Russia